CLINICAL TRIAL: NCT06041906
Title: International Registry of Congenital Portosystemic Shunts (IRCPSS) - A Multi-centre, Retrospective and Prospective Registry of Neonates, Children and Adults With Congenital Portosystemic Shunts
Brief Title: International Registry of Congenital Portosystemic Shunt (IRCPSS)
Acronym: IRCPSS
Status: Enrolling by invitation | Type: Observational
Sponsor: Prof. Valérie Mc Lin (Other)
Collaborators: European Society of Pediatric Gastroenterology, Hepatology and Nutrition (Other); European Association for the Study of the Liver (EASL) (Unknown); Fondation Andrea Ferrari (Unknown)
Responsible Party: Sponsor-Investigator, Prof. Valérie Mc Lin, Prof. Dr. med., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2018-00413
Record Dates: First submitted 2023-09-11; First posted 2023-09-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2024-12

CONDITIONS: Congenital Portosystemic Shunt; CPSS (Congenital Portosystemic Shunt)
Keywords: shunt; portosystemic; portasystemic; porto-systemic; porta-systemic; registry; liver; rare disease; Abernethy malformation; vascular malformation; Hypertension, Pulmonary; Hepatopulmonary Syndrome; Liver Neoplasms; hyperinsulinemic; hypoglycemia; hyperinsulinism; Insulin resistance; hyperandrogenism; Hepatic Encephalopathy; Hyperammonemia
MeSH Terms: conditions — Congenital Portosystemic Shunt; Rare Diseases; Vascular Malformations; Hypertension, Pulmonary; Hepatopulmonary Syndrome; Liver Neoplasms; Hypoglycemia; Hyperinsulinism; Insulin Resistance; Hyperandrogenism; Hepatic Encephalopathy; Hyperammonemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Neonate, Children, Adult with CPSS
  Interventions: Procedure: Shunt Closure

INTERVENTIONS:
Procedure: Shunt Closure — Consist in spontaneous, surgical or interventional closure of the shunt. Depending on context, surgical intervention may also be transplantation.

SUMMARY:
Congenital Portosystemic Shunt (CPSS) is a rare condition important by the multiplicity and severity of associated complications.

CPSS is venous anomaly in which blood coming from the intestines only partially passes through the liver.

This leads to the accumulation of potentially toxic factors that cause systemic effects.

Complications vary among the individuals, and currently, it is challenging to predict which individuals will develop severe complications.

The IRCPSS registry is established with the aim of centralizing detailed clinical follow-up and biological information from participants around the world who suffer from Congenital Portosystemic Shunt (CPSS). A multidisciplinary consortium of experts is collaborating to enhance our understanding of the prevalence, natural history, individual risks, and physiopathology of the disease through the IRCPSS registry.

ELIGIBILITY:
Inclusion Criteria:

Individual with CPSS

Exclusion Criteria:

Secondary shunt without evidence of congenital shunt

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: neonates; children; adults
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2026-10-26 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Numbers of patients with spontaneous shunt closure | 3; 6; 12; 24 months
Number of patients developing one or more complications | 5; 10; 20 years
Number of patients undergoing preemptive closure | 6; 12; 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Valérie A Mc Lin, Prof. Dr. med., Study Director — University Hospital, Geneva
Locations (26):
- United States (2):
  - Yale University School of Medicine, New Haven, Connecticut
  - Lurie Children's Hospital, Chicago, Illinois
- Royal Children's Hospital Melbourne, Parkville, Victoria, Australia
- Universitary Clinics Saint-Luc, UCL, Brussels, Belgium
- The Hospital for Sick Children, Toronto, Ontario, Canada
- France (3):
  - Beaujon University Hospital, Clichy
  - Hôpital Bicêtre-Hôpitaux Universitaires Paris-Sud- Assistance Publique Hôpitaux de Paris., Le Kremlin-Bicêtre
  - Hôpital Necker, Paris
- Germany (3):
  - Hannover Medical School, Hanover
  - Haunersche Kinderklinik - LMU Munich, Munich
  - University of Tuebingen, Tübingen
- First Department of Pediatrics, Semmelweis University, Budapest, Hungary
- India (2):
  - Amrita institute of Medical Sciences, Kochi, Kerala
  - Department of Pediatric Hepatology Institute of Liver and Biliary Sciences, New Delhi
- Schneider Children's Medical Center of Israel, Petach Tikvah, Israel
- Italy (3):
  - Papa Giovanni XXIII Hospital, Bergamo
  - Children's Hospital Santobono, Naples
  - Istituto di Ricovero e Cura a Carattere Scientifico (ISMETT), Palermo
- National Center for Child Health and Development, Tokyo, Japan
- Netherlands (2):
  - Academic Medical Centre, Amsterdam
  - University Medical Center Groningen, Groningen
- Hospital Clínic de Barcelona, Barcelona, Spain
- Hôpitaux Universitaires de Geneve (HUG), Geneva, Canton of Geneva, Switzerland
- Gazi University, Faculty of Medicine, Yenimahalle, Ankara, Turkey (Türkiye)
- United Kingdom (2):
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Children and Young People, Edinburgh

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Hanquinet S, Morice C, Courvoisier DS, Cousin V, Anooshiravani M, Merlini L, McLin VA. Globus pallidus MR signal abnormalities in children with chronic liver disease and/or porto-systemic shunting. Eur Radiol. 2017 Oct;27(10):4064-4071. doi: 10.1007/s00330-017-4808-x. Epub 2017 Apr 6. PMID 28386718
- [Background] Cudalbu C, McLin VA, Lei H, Duarte JM, Rougemont AL, Oldani G, Terraz S, Toso C, Gruetter R. The C57BL/6J mouse exhibits sporadic congenital portosystemic shunts. PLoS One. 2013 Jul 23;8(7):e69782. doi: 10.1371/journal.pone.0069782. Print 2013. PMID 23936100
- [Background] Joye R, Lador F, Aggoun Y, Farhat N, Wacker J, Wildhaber BE, Vallee JP, Hachulla AL, McLin VA, Beghetti M. Outcome of paediatric portopulmonary hypertension in the modern management era: A case report of 6 patients. J Hepatol. 2021 Mar;74(3):742-747. doi: 10.1016/j.jhep.2020.11.039. Epub 2020 Dec 1. PMID 33276028
- [Background] McLin V, Beghetti M, D'Antiga L, Franchi-Abella S; International Registry of Congenital Porto-Systemic Shunts (IRCPSS). Current Quandaries in the Management of Congenital Portosystemic Shunts. Liver Transpl. 2021 Aug;27(8):1212-1213. doi: 10.1002/lt.26055. Epub 2021 Jul 20. No abstract available. PMID 33749116
- [Background] Korff S, Mostaguir K, Beghetti M, D'Antiga L, Debray D, Franchi-Abella S, Gonzales E, Guerin F, Hachulla AL, Lambert V, Makrythanasis P, Roduit N, Savale L, Senat MV, Spaltenstein J, van Steenbeek F, Wildhaber BE, Zwahlen M, McLin VA. International registry of congenital porto-systemic shunts: a multi-centre, retrospective and prospective registry of neonates, children and adults with congenital porto-systemic shunts. Orphanet J Rare Dis. 2022 Jul 19;17(1):284. doi: 10.1186/s13023-022-02412-8. PMID 35854389
- [Background] Lambert V, Ladarre D, Fortas F, Durand P, Herve P, Gonzales E, Guerin F, Savale L, McLin VA, Ackermann O, Franchi-Abella S; International Registry of Congenital Portosystemic Shunts (IRCPSS). Cardiovascular disorders in patients with congenital portosystemic shunts: 23 years of experience in a tertiary referral centre. Arch Cardiovasc Dis. 2021 Mar;114(3):221-231. doi: 10.1016/j.acvd.2020.10.003. Epub 2020 Dec 3. PMID 33281106
- [Background] McLin VA, D'Antiga L. The current pediatric perspective on type B and C hepatic encephalopathy. Anal Biochem. 2022 Apr 15;643:114576. doi: 10.1016/j.ab.2022.114576. Epub 2022 Jan 29. PMID 35104444
- [Background] McLin VA, Franchi Abella S, Debray D, Guerin F, Beghetti M, Savale L, Wildhaber BE, Gonzales E; Members of the International Registry of Congenital Porto-Systemic Shunts. Congenital Portosystemic Shunts: Current Diagnosis and Management. J Pediatr Gastroenterol Nutr. 2019 May;68(5):615-622. doi: 10.1097/MPG.0000000000002263. PMID 30628988
- [Background] Bahadori A, Kuhlmann B, Debray D, Franchi-Abella S, Wacker J, Beghetti M, Wildhaber BE, McLin VA, On Behalf Of The Ircpss. Presentation of Congenital Portosystemic Shunts in Children. Children (Basel). 2022 Feb 11;9(2):243. doi: 10.3390/children9020243. PMID 35204963
- [Background] Guerin F, Franchi Abella S, McLin V, Ackermann O, Girard M, Cervoni JP, Savale L, Hernandez-Gea V, Valla D, Hillaire S, Dutheil D, Bureau C, Gonzales E, Plessier A. Congenital portosystemic shunts: Vascular liver diseases: Position papers from the francophone network for vascular liver diseases, the French Association for the Study of the Liver (AFEF), and ERN-rare liver. Clin Res Hepatol Gastroenterol. 2020 Sep;44(4):452-459. doi: 10.1016/j.clinre.2020.03.004. Epub 2020 Apr 9. No abstract available. PMID 32279979
- [Background] Rock NM, Beghetti M, Tissot C, Willi JP, Bouhabib M, McLin VA, Maggio ABR. Reliable Detection of Intrapulmonary Shunts Using Contrast-Enhanced Echocardiography in Children With Portal Hypertension or Portosystemic Shunt. J Pediatr Gastroenterol Nutr. 2021 Jul 1;73(1):73-79. doi: 10.1097/MPG.0000000000003079. PMID 33605662
- See also: International Registry of Congenital Portosystemic Shunts website, for patients and professionals — https://ircpss.com/